CLINICAL TRIAL: NCT03886558
Title: Effects of a Long Term Multicomponent Intervention Program on a Group of Nonagenarians
Brief Title: Multicomponent Program on a Group of Nonagenarians
Acronym: ELTGN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, José M. Cancela, PhD, University of Vigo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IPVC 2017-123
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Quality of Life; Healthy; Aging; Physical Activity
Keywords: exercise; longevity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: A multicomponent intervention program was developed consisting of two 60-minute sessions per week, held on non-consecutive days, for a period of 8 months. The sessions consisted of a warm-up phase (10') in which individuals performed joint mobility exercises and walked at a rate of 3 km/h. Afterwards, muscular strength work was carried out on the upper and lower limbs, including calisthenic exercises, and the use of dumbbells or medicine balls (1-3kg). Generally, the exercises were organized in two sets of 10-15 repetitions, resting for two minutes between sets. Communal ball games and relay games were then practiced (over a distance of 30 meters). Finally, 10 minutes were devoted to relaxation and stretching exercises. multicomponent intervention program was designed and monitored by a specialist in gerontogymnastics.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Institution Group (n=14) (Experimental): A multicomponent intervention program was developed consisting of two 60-minute sessions per week, held on non-consecutive days, for a period of 8 months. The sessions consisted of a warm-up phase (10') in which individuals performed joint mobility exercises and walked at a rate of 3 km/h. Afterwards, muscular strength work was carried out on the upper and lower limbs, including calisthenic exercises, and the use of dumbbells or medicine balls (1-3kg). Generally, the exercises were organized in two sets of 10-15 repetitions, resting for two minutes between sets. Communal ball games and relay games were then practiced (over a distance of 30 meters). Finally, 10 minutes were devoted to relaxation and stretching exercises. multicomponent intervention program was designed and monitored by a specialist in gerontogymnastics.
  Interventions: Other: A multicomponent intervention program was developed consisting of two 60-minute sessions per week, held on non-consecutive days, for a period of 8 months.
- Community Group (n=16) (Experimental): A multicomponent intervention program was developed consisting of two 60-minute sessions per week, held on non-consecutive days, for a period of 8 months. The sessions consisted of a warm-up phase (10') in which individuals performed joint mobility exercises and walked at a rate of 3 km/h. Afterwards, muscular strength work was carried out on the upper and lower limbs, including calisthenic exercises, and the use of dumbbells or medicine balls (1-3kg). Generally, the exercises were organized in two sets of 10-15 repetitions, resting for two minutes between sets. Communal ball games and relay games were then practiced (over a distance of 30 meters). Finally, 10 minutes were devoted to relaxation and stretching exercises. multicomponent intervention program was designed and monitored by a specialist in gerontogymnastics.
  Interventions: Other: A multicomponent intervention program was developed consisting of two 60-minute sessions per week, held on non-consecutive days, for a period of 8 months.

INTERVENTIONS:
Other: A multicomponent intervention program was developed consisting of two 60-minute sessions per week, held on non-consecutive days, for a period of 8 months. — The sessions consisted of a warm-up phase (10') in which individuals performed joint mobility exercises and walked at a rate of 3 km/h. Afterwards, muscular strength work was carried out on the upper and lower limbs, including calisthenic exercises, and the use of dumbbells or medicine balls (1-3kg). Generally, the exercises were organized in two sets of 10-15 repetitions, resting for two minutes between sets. Communal ball games and relay games were then practiced (over a distance of 30 meters). Finally, 10 minutes were devoted to relaxation and stretching exercises. multicomponent intervention program was designed and monitored by a specialist in gerontogymnastics.

SUMMARY:
Introduction The promotion of physical activity among older adults is considered to be one of the main actions that can result in more successful aging. Currently, there are few studies focusing on the effects of long-duration physical activity interventions in older adults. Thus, the purpose of the following study was to analyze the effects of an 8-month multicomponent intervention program on cardiorespiratory capacity, body composition, and strength in a group of nonagenarians. A secondary objective was to determine if the impact of the program differed according to the participants' way of life (institutionalized vs. community dwelling).

Methods Participants Participants in this research represent a subset from an ongoing study aimed at collecting baseline and follow-up data over three years, to evaluate the health-related changes observed in a cohort of older adults f The present research was carried out on the basis of data obtained from the individuals in this sample who participated in a multicomponent intervention program offered to the inhabitants of the said region and who met the following inclusion criteria: a) being ninety years of age or older; and b) holding a medical certificate confirming their suitability for sport. The exclusion criteria were a) lack of independent ambulation (walking with an assistive device); b) recent upper or lower limb injuries; c) neurological or orthopedic diagnosis in upper or lower-extremities.

Intervention A multicomponent intervention program was developed consisting of two 60-minute sessions per week, held on non-consecutive days, for a period of 8 months. The sessions consisted of a warm-up phase (10') in which individuals performed joint mobility exercises and walked at a rate of 3 km/h. Afterwards, muscular strength work was carried out on the upper and lower limbs, including calisthenic exercises, and the use of dumbbells or medicine balls (1-3kg). Generally, the exercises were organized in two sets of 10-15 repetitions, resting for two minutes between sets. Communal ball games and relay games were then practiced (over a distance of 30 meters). Finally, 10 minutes were devoted to relaxation and stretching exercises. multicomponent intervention program was designed and monitored by a specialist in gerontogymnastics.

Evaluations Two weeks before the start and after the end of the exercise program, a series of assessments were carried out, which were monitored by specialists in physical exercise and sport, who did not know whether those evaluated were institutionalized or not.

Body composition Weight was measured to the nearest 0.1 kg using a Tefal digital scale (type PP1200VO) with the participants wearing light clothing and no shoes. Height was measured to the nearest millimeter with a field stadiometer (Seca 220). The body mass index (BMI) was calculated taking the body weight in kilograms and dividing it by the height in meters squared (BMI: kg/m2).

Densitometry Bone mineral density content (BMD) of the femoral neck was measured using a dual energy X-ray absorptiometry (DEXA) machine (Hologic QDR 1000®), which reported BMD in grams per square centimeter (g/cm2). This method was used to ensure better reproducibility, a lower radiation dose and better image resolution (Watts 2004). The minimum significant alteration, with a 95% confidence interval, was 4.7%.

Muscular strength Upper limb muscle strength was assessed with the Handgrip Test (HG) on the right hand using a dynamometer (SH5001, SAEHAN Corporation, South Korea). For each measurement, patients were asked to perform their maximum voluntary contraction for 5s. Each measurement was repeated three times with patients resting for 30s between trials. The best performance was recorded for further analysis. Lower limb muscle strength was assessed with the Isometric Knee Extension Test (KNEE), performed three times on the right leg with participants seated on a custom-built chair with a load cell (Vetek VZ101BS, Vaddo, Sweden). For each measurement, participants were asked to perform their maximum voluntary contraction for 5 s. The test was repeated 3 times and participants rested for 2 min between trials. The best performance from the three trials was considered for further analysis.

Cardiorespiratory fitness In order to assess the effect of the program on the participants' cardiorespiratory fitness, the six-minute walk test (6MWT), was performed, following standard procedure. The subjects were instructed to walk at their own pace from one end to the other of a 100-foot-long measured distance in an enclosed, level, corridor, and to cover as much ground as possible in 6 min. They were allowed to stop and rest during the test, but were instructed to resume walking as soon as they felt able to do so.

ELIGIBILITY:
Inclusion Criteria:

1. being ninety years of age or older;
2. holding a medical certificate confirming their suitability for sport.

Exclusion Criteria:

1. lack of independent ambulation (walking with an assistive device);
2. recent upper or lower limb injuries;
3. neurological or orthopedic diagnosis in upper or lower-extremities

Min Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Body composition | 32 weeks
  Weight was measured to the nearest 0.1 kg using a Tefal digital scale (type PP1200VO) with the participants wearing light clothing and no shoes. Height was measured to the nearest millimeter with a field stadiometer (Seca 220). The body mass index (BMI) was calculated taking the body weight in kilograms and dividing it by the height in meters squared (BMI: kg/m2).
Densitometry | 32 weeks
  Bone mineral density content (BMD) of the femoral neck was measured using a dual energy X-ray absorptiometry (DEXA) machine (Hologic QDR 1000®), which reported BMD in grams per square centimeter (g/cm2). This method was used to ensure better reproducibility, a lower radiation dose and better image resolution (Watts 2004). The minimum significant alteration, with a 95% confidence interval, was 4.7%.
Muscular strength | 32 weeks
  Upper limb muscle strength was assessed with the Handgrip Test (HG) on the right hand using a dynamometer (SH5001, SAEHAN Corporation, South Korea). For each measurement, patients were asked to perform their maximum voluntary contraction for 5s. Each measurement was repeated three times with patients resting for 30s between trials. The best performance was recorded for further analysis. Lower limb muscle strength was assessed with the Isometric Knee Extension Test (KNEE), performed three times on the right leg with participants seated on a custom-built chair with a load cell (Vetek VZ101BS, Vaddo, Sweden). For each measurement, participants were asked to perform their maximum voluntary contraction for 5 s. The test was repeated 3 times and participants rested for 2 min between trials. The best performance from the three trials was considered for further analysis.
Cardiorespiratory fitness | 32 weeks
  In order to assess the effect of the program on the participants' cardiorespiratory fitness, the six-minute walk test (6MWT), was performed, following standard procedure. The subjects were instructed to walk at their own pace from one end to the other of a 100-foot-long measured distance in an enclosed, level, corridor, and to cover as much ground as possible in 6 min. They were allowed to stop and rest during the test, but were instructed to resume walking as soon as they felt able to do so.

CONTACTS AND LOCATIONS:
Locations (1):
- Univerity of Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Undecided